CLINICAL TRIAL: NCT00911001
Title: Compliance and Treatment Satisfaction in Prophylaxis of Postsurgical Thromboembolism
Brief Title: SALTO - Epidemiological Study on Compliance and Treatment Satisfaction
Acronym: SALTO
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14343; NN0811ES
Record Dates: First submitted 2009-05-27; First posted 2009-06-01 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Thromboembolism
Keywords: Arthroplasty; Antithrombotic prophylaxis treatment; Replacement; Knee
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Behavioral: No Drug

INTERVENTIONS:
Behavioral: No Drug — Patients in daily life clinical treatment receiving pharmacological agents to prevent VTE.

SUMMARY:
Patients that are on total knee/hip replacement initiate prophylaxis treatment on the hospital ground. Once they leave the hospital, as outpatients they continue with the treatment at least during two consecutive weeks. Patients will be instructed to follow treatment recommendations (either LMWH or oral treatment, at physician discretion) and to come back to the surgeon after that period. At that visit, the Treatment Satisfaction Questionaire with Medication (TSQM) test as well as the Moriski-Green Questionaire (measures compliance with medication) will be answer by the patient. TSQM is an self administered validated scale (validated also in spanish) that measures in a generic way the treatment satisfaction to a treatment. Morinski-Green test will be used to measure the compliance degree on medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients in antithrombotic prophylaxis treatment after total knee/hip replacement. This is an epidemiological study where the patients to be included will be those that are treated with antithrombotics as out-patients in real life conditions.

Exclusion Criteria:

* Patients who has been previously treated with injectable antithrombotic treatments.
* Diabetic patients treated with insulin.
* Patients who do not sign Informed Consent Form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in antithrombotic prophylaxis treatment after total knee/hip replacement
Sampling Method: Non-Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2008-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To measure the Treatment Satisfaction with medication through the self administered scale TSQM. | 2 weeks

SECONDARY OUTCOMES:
To measure compliance with medication and the relationship with satisfaction through the Moriski-Green Questionaire | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Spain